CLINICAL TRIAL: NCT05990062
Title: The Advancement of a New Variable-Compliance Socket and Frame System for Transradial Amputees to Optimize Socket Fit and Upper Limb Function
Brief Title: Improving Prosthetic Arms for Amputee: A Better Fit and More Functionality
Acronym: KSH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Stumpworx LLC (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A4257-R
Record Dates: First submitted 2023-07-18; First posted 2023-08-14 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Amputation, Surgical
Keywords: function; breathability; comfort; transradial

STUDY DESIGN:
Intervention Model Description: The protocol consists of three phases with iterative design and development process involving input from Veterans with disabilities at various stages. In addition, 5 certified Prosthetists with at least five years of experience working with Veterans with transradial arm amputations will also be recruited to provide guidance and to assist with the design and development of the K-Socket Harness (KSH).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Verify performance gains for the innovative KSH system that can be delivered to Veterans. The new de (Experimental): The investigators will perform several functional tests of the both the KSH system and the standard of care prosthesis: tensile static load bearing capacity before failure, test rowing ergometer 10-minute test before failure measured using strokes per minute, power in Watts, distance in meters, maximal force, and time before failure, range of motion in flexion/extension, and donning/doffing time.
  Interventions: Device: K-Socket-Harness
- Verify functionality of the KSH system through testing with end-users. (Experimental): The investigators will use System Usability Scale (SUS) to assess high usability with setup and operation of the device. The investigators will assess Comfort Scores (SCS), evaluate weight and correlate it with user satisfaction. The investigators will report selection outcome between new design and current design. The investigators will asses 1) functional status, (2) health- related quality of life, and (3) satisfaction with services and (4) device scores through the Orthotics and Prosthetics User Survey (OPUS).
  Interventions: Device: K-Socket-Harness

INTERVENTIONS:
Device: K-Socket-Harness — A transradial socket and harness design that offers a hybrid polymer and textile-based design derived from advanced athletic shoe technology. The KSH integrated socket, frame, and wrist, the "variable compliance prosthetic socket with breathable matrix," creates a dynamic and secure attachment with a combination of two lacing systems. The lacing systems lengthen and shorten six flexible hinges at the elbow, maintaining a secure attachment throughout the range of motion and accounting for volume changes in the soft tissue of the elbow that would otherwise restrict range of motion or cause the socket to separate from the residual limb.
  Other Names: KSH System

SUMMARY:
This research and development will improve upon and investigate the potential validity of an innovative new transradial socket and harness design (the KSH system) that offers an alternative to standard hard sockets and rubber liners with a hybrid polymer and textile-based design derived from advanced athletic shoe technology. The project consists of designing, custom fitting and evaluating the function and comfort of the this new novel system. The study will take place in 3 phases; Phase 1, five experienced Veterans with transradial arm amputations will be recruited to provide guidance and to assist with the design and development. Experienced end-user Veterans and Clinical staff will work together to assist with design, develop the fitting process and working with engineers on the design of a completely digital fitting device for measuring the residual limb and locating bony prominences of the limb to inform the socket design. Phase 2, testing and assessment, the design and process validation will take place with the five Veteran upper transradial arm amputees Phase 3, an additional 20 Veterans with transradial arm amputations will be recruited and fit with the KSH system and undergo a series of evaluative tests. Veterans will perform a series of static and dynamic tasks to evaluate function, comfort and load bearing failure. The primary goal of this study is to improve upon the current preliminary prototype and to test it with a broader population of potential users to help advance the engineering and design, and to learn the potential to fit a range of Veterans with transradial amputations.

DETAILED DESCRIPTION:
Acceptance of prosthetic arms has long been a problem for clinical prosthetics, and recent studies indicate that recent advancements have done little to improve usage. Objections related to the fit and comfort of prosthetic arms remain the main reasons cited for the disuse of the devices, numbering nine of the top ten reasons cited for abandonment in a survey study. By addressing the literal point of pain for these users, the investigators hope to increase use and acceptance, allowing existing devices to have more positive impact on Veterans' lives. The breathability of composite sockets has been an acknowledged problem nearly since their development by the VA in the 1940s. Indeed, while the VA successfully developed a breathable composite socket very early on, it was quickly abandoned after it was discovered that the breathable composite recreated the problems with odor and cleanliness with leather sockets that the composites had been developed to solve. Industry leader Otto Bock discovered the same thing when it developed a porous silicone liner decades later. While VA and civilian providers were successful in replacing leather sockets with composites through the innovations in composites and other materials following World War II. Prosthetic clinics used to employ leatherworkers skilled in the art of making custom sockets and braces out of these traditional materials, but these services have disappeared along with the Veterans demanding them, and the workers capable of delivering them. By taking advantage of the benefits of the advanced materials and construction techniques that have replaced leather in the athletic shoe industry over the last seventy-five years, the investigators hope to restore much of the comfort and fit of these extinct socket designs, while at the same time delivering the improvements that have been delivered by the athletic shoe industry and advances in design and manufacturing over the same period. Lim design is working on a textile based prosthetic socket; however, the approach differs from the investigators': 1) The Lim design is not intended or currently suitable for upper limbs; 2) While a textile design, the Lim design cannot dynamically change in volume through the range of motion and constrains motion similar to any other socket once it has been adjusted; 3) The textile design of the Lim socket is nether breathable nor wicking and is designed to be used with silicone and/or gel liners, hence suffers from the same deficiencies with respect to heat and moisture management as traditional sockets. Lim Innovations and Ossur have publicly stated that they do not intend to pursue further innovations in the upper limb market. These frank admissions make it clear that the development of orphan devices for Veterans, must become the responsibility of the VA, whose goals for serving Veterans are sometimes in contrast with and not limited to the constraints of large and profitable markets. VA in collaboration with small companies can help fill this much needed void for innovation. VA has shown leadership in related domains with the research and design for ultralight wheelchairs, alternative controls for powered wheelchairs, and adaptive sports and recreation equipment, all of which eventually assisted the broader populations of Americans with disabilities. Harness discomfort is just as detrimental to acceptance as poor socket-body interface and can lead to contralateral damage to the axilla. Indeed, one recent study concluded that there was no acceptable level of force at which a body powered prosthesis could be operated pain and fatigue free with a traditional harness. While the conclusions of this study obviously contradict the staying power of the body powered prosthesis and harness system accepted by more than 90 per cent of the roughly half of users who accept a prosthesis at all, it does indicate that there is substantial improvement to be made in harnessing that could significantly improve both acceptance and comfort of the users who have been willing to tolerate the uncomfortable standard of care that has seen slow progress for decades.

Study Objectives and Hypothesis:

Specific Aim 1: Improve and develop the design and systems for fitting an innovative new transradial suspension design based on currently available technology used in athletic shoe construction.

* Design Criteria 1a: Optimize CAD documentation by revising and translating the current Autodesk Fusion 360 design to SolidWorks, aiding customization and improving design for manufacture.
* Design Criteria 1b: Verify that the currently Direct Metal Laser Sintered (DMLS) printed wrist and quick release can be efficiently and effectively CNC machined.
* Design Criteria 1c: Create fixturing and finalize CNC programming for manufacture, including the specification of manufacturing tolerances to ensure proper fit of components.
* Design Criteria 1e: Verify forearm and elbow counter parts-currently printed in Multijet Fusion (MJF)-in Selective Laser Sintering (SLS) or Fused Deposition or Fused Filament (FDM/FFF) Nylon material.
* Design Criteria 1f: Automate adaptation of the design through plugin and API development.
* Design Criteria 1g: Optimize production of 2D textile patterns with, for example, ExactFlat.
* Design Criteria 1h: Design a digital or Brannock-like fitting device for measuring the residual limb and locating bony prominences of the limb to inform the socket design.
* Design Criteria 1i: Design the device to weigh less than 2-pounds total weight. Jon is a 50-year-old Veteran with a transradial arm amputation. He has had multiple carpal tunnel release surgeries on his remaining hand. An inconsistent but long-term user of prostheses, Jon settled on body-powered arms after extensive trials of myoelectric prostheses at Walter Reed immediately following his injury in Iraq in 2005, primarily because of the discomfort and lack of range of motion in the socket. He uses them mostly for true bimanual tasks, including bicycle riding, hunting, shotgun sports, and home improvement. Jon was not selected for a trial of the DEKA arm in 2018, and instead received a Bebionic hand and hard self-suspended socket from the VA. This arm was quickly rejected: it was heavy, incapable, uncomfortable, and restrictive. Blistering and irritation to Jon's arm from sweating and friction in a silicone lined carbon fiber vacuum socket.

Specific Aim 2: Verify performance gains for the innovative KSH system that can be delivered to Veterans. The new design is expected to significantly exceed the performance of the standard-of-care prosthesis in quantitative measures.

* Hypothesis 2a (H2a): That the improved KSH will provide a higher tensile static load bearing capacity before failure than the current standard-of-care prosthesis.
* Hypothesis 2b (H2b): That the improved KSH will provide greater tensile loads in a dynamic environment. The KSH system will allow users to perform better on a rowing ergometer 10-minute test before failure than the current standard-of-care prosthesis, as measured using strokes per minute, power in Watts, distance in meters, maximal force, and time before failure.
* Hypothesis 2c (H2c): The improved KSH will provide a greater range of motion in flexion/extension than the current standard-of-care prosthesis.
* Hypothesis 2d (H3d): Participants will require less time for donning/doffing the KSH than their current standard-of-care prosthesis.

Specific Aim 3: Verify functionality of the KSH system through testing with end-users.

* Hypothesis 3a (H3a): Participants will report high usability with setup and operation of the device (>80 on the System Usability Scale (SUS)).
* Hypothesis 3b (H3b): Participants will report significantly higher Socket Comfort Scores (SCS) with the KSH than their current standard-of-care prosthesis.
* Hypothesis 3c (H3c): Lower weight will correlate with greater user satisfaction, and the KSH will be statistically and clinically significantly lighter than participants' current devices.
* Hypothesis 3d (H3d): Participants will report that they would switch to the new design or have an additional prosthesis with the new design.
* Hypothesis 3e (H3e): Participants will report significantly higher Orthotics and Prosthetics User Survey (OPUS) scores with the KSH than their current standard-of-care prosthesis.

Relevance to Veterans: According to the DoD/VA Extremity Amputation Center of Excellence there were about 3,000 Veterans with transradial amputations enrolled for VA Healthcare in FY21, out of about 62,000 Veterans with limb amputations enrolled for VA healthcare. Veterans with arm amputations from Post-911 conflicts number just over 200, and because the total number of Veterans missing arms is demographically small, this very fact has severely limited innovation in the field of prosthetic arms. Those missing at least all five fingers of a hand are among the VA's most significantly disabled Veterans, rated at 80 per cent disabled alone for the loss of a dominant hand. Many arm amputees are eligible for Special Monthly Compensation as well as vehicle and housing modifications, reflecting the degree to which these Veterans' lives are impacted by the impairment. Indeed, even among the civilian population, arm amputation is rare enough to easily meet the FDA's medical orphan criteria of fewer than 200,000 patients, though the FDA's orphan drug law specifically excludes medical devices, and the FDA has a lower device threshold of 8,000 patients, further limiting innovation. The NIH's Genetic and Rare Diseases Information Center (GARD) lists limb absence as a rare birth condition but doesn't mention the same disability acquired by trauma or through other diseases, such as cancer, which is the second most common cause despite the small total number from all causes. While the subject design can be extended to other levels of amputation, this study will focus on transradial, or below elbow amputees. This population represents approximately seventy-five per cent of the VA population of Veterans with arm amputations, a subset that is also much more likely to successfully wear a prosthetic arm. Over 90% of these users choose body powered. The design could be extended to other Veteran populations, including people with lower-limb amputations and other levels of amputation, potentially increasing the benefit by offering the same benefits to those Veterans. By targeting the portion of an orphan population that is already more likely to use the device for which improvement is sought, and by targeting the concerns that are most likely to lead to abandonment, this research stands to increase acceptance and therefore access to activities of daily living, employment and recreation that can improve quality of life for some of the VA's most impaired patients. Success could then also be translated to larger populations with similar needs. The proposed design is intended to address more than half the total population of Veterans with upper limb amputations and could with additional research and development be designed in the future for other levels of amputation, including lower limb and myoelectric upper limb use.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transradial arm amputation
* Possession of a functioning and wearable previously fit prosthetic arm of any type
* Residual limb length of at least 4 inches from the lateral epicondyle to the distal tip
* Residual limb length less than or equal to that allowing a clearance of 1.5 inches from a fitted wrist
* Must have at least 5-years of prosthetic use experience (For Phase 1 & 2)
* Must have at least 1-year of prosthetic use experience (For Phase 3 only)

Exclusion Criteria:

* Current open sores or incisions, Heterotopic ossification (HO), traumatic neuromas, or any other condition preventing the wearing of a prosthetic socket
* Residual limb length less than 4 inches
* Residual limb length greater than that allowing 1.5 inches clearance from a fitted wrist.

The investigators will make every effort to recruit Veterans. If its found that it is not possible to recruit enough Veterans, the investigators will perform a non-Veteran amendment to this protocol.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Static tensile load bearing capacity to reach a 50-pound load on an industrial scale | 20 minutes
  We will test tensile static load bearing capacity up to a 50 -pound load or to failure. The Veteran will stand safely on an industrial scale with the arm extended at their side and weight will be added to the distal end of the prosthesis until the goal is met or the prosthesis fails. We will perform the task on both the KSH socket and the standard socket.
Elbow range of motion in flexion/extension | 30 minutes
  We will measure range of motion (in degrees) in flexion/extension with a standard goniometer. We will perform the task on both the KSH socket and the standard socket.
Donning/doffing prosthesis | 30 minutes
  We will record the time it takes to donn/doff each prosthesis for both the KSH socket and the standard socket.
Power in Watts generated on rowing machine | 10 minutes
  We will test tensile loads in a dynamic environment before failure. We will test the performance on a rowing ergometer 10-minute test before failure, as measured using power in Watts. We will perform the task on both the KSH socket and the standard socket.
Strokes per 10-minute period | 10 minutes
  We will test tensile loads in a dynamic environment before failure. We will test the performance on a rowing ergometer 10-minute test before failure, as measured using strokes per minute. We will perform the task on both the KSH socket and the standard socket.
Distance rowed in meters | 10 minutes
  We will test tensile loads in a dynamic environment before failure. We will test the performance on a rowing ergometer 10-minute test measuring distance in meters before failure or to time expiration. We will perform the task on both the KSH socket and the standard socket.
Maximal force before failure | 10 minutes
  We will test tensile loads in a dynamic environment before failure. We will test the performance on a rowing ergometer 10-minute test measuring maximal force (Newton) before failure. We will perform the task on both the KSH socket and the standard socket.
Total time before failure | 10 minutes
  We will test tensile loads in a dynamic environment before failure. We will test the performance on a rowing ergometer 10-minute test recording the time (in minutes and seconds) before failure. We will perform the task on both the KSH socket and the standard socket.

SECONDARY OUTCOMES:
Usability of prosthesis using the System Usability Score (SUS) on scale from 0-100 | 15 minutes
  Participants will report usability with setup and operation of the device from ten questions using a five point Likert scale. The higher the score, the more usable (user friendly) the device is rated by the Veteran. We would like the KSH system to score >80 on the System Usability Scale (SUS)).
Socket Comfort Scores (SCS) on a scale from 0-10 | 30 minutes
  Participants will report Socket Comfort Scores (SCS) after wearing and testing of the devices for both with the KSH and current standard-of-care prosthesis by using an 11 point scale, (0-10) Zero being the most uncomfortable socket fit you can image, and 10 being the most comfortable socket fit.
Weight of device in pounds | 30 minutes
  We will correlate the weight of the prosthesis in pounds with user satisfaction of both the KSH device and the participants' current device.
Participant preference | 10 minutes
  We will ask the participant which device design they prefer to use.
Orthotics and Prosthetics User Survey (OPUS) | 1 hour
  We will ask the participant to complete the questionnaire focusing on five modules; lower and upper extremity functional status (LEFS and UEFS), client satisfaction with device and services (CSD and CSS), and the health related quality of life (HRQoL) Scores are based on a 100 point scale. The higher the score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Rory A Cooper, PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Any information obtained from this study will be treated as confidential and will be safeguarded in accordance with the HIPAA privacy and security regulations. Research records may be released or disclosed if required by federal law. Records will be coded by assigning a case number and the information linking the case number to the subject's identity will be stored electronically on the VAPHS network. Any protected health information (PHI) stored electronically is in compliance with the HIPAA security rule. Study subjects will not be specifically identified in any publication of research results. Paper source documents of the coded research records will be kept in file cabinets within a locked file room. Any records which contain direct subject identifiers will be stored separately, with a different identification code, in a locked file cabinet within a locked file room. Records will be maintained in accordance with the Veterans Health Administration (VHA) Records Control Schedule.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data sharing will begin upon the start of enrolling the first subject (10/1/2024) and end at the completion of the study (9/30/2028).

REFERENCES:
- [Background] Salminger S, Stino H, Pichler LH, Gstoettner C, Sturma A, Mayer JA, Szivak M, Aszmann OC. Current rates of prosthetic usage in upper-limb amputees - have innovations had an impact on device acceptance? Disabil Rehabil. 2022 Jul;44(14):3708-3713. doi: 10.1080/09638288.2020.1866684. Epub 2020 Dec 30. PMID 33377803
- [Background] Biddiss E, Chau T. Upper-limb prosthetics: critical factors in device abandonment. Am J Phys Med Rehabil. 2007 Dec;86(12):977-87. doi: 10.1097/PHM.0b013e3181587f6c. PMID 18090439
- [Background] Hichert M, Vardy AN, Plettenburg D. Fatigue-free operation of most body-powered prostheses not feasible for majority of users with trans-radial deficiency. Prosthet Orthot Int. 2018 Feb;42(1):84-92. doi: 10.1177/0309364617708651. Epub 2017 Jun 16. PMID 28621577
- [Background] Hanspal RS, Fisher K, Nieveen R. Prosthetic socket fit comfort score. Disabil Rehabil. 2003 Nov 18;25(22):1278-80. doi: 10.1080/09638280310001603983. PMID 14617445
- [Background] Heinemann AW, Bode RK, O'Reilly C. Development and measurement properties of the Orthotics and Prosthetics Users' Survey (OPUS): a comprehensive set of clinical outcome instruments. Prosthet Orthot Int. 2003 Dec;27(3):191-206. doi: 10.1080/03093640308726682. PMID 14727700
- [Background] Dillingham TR, Pezzin LE, MacKenzie EJ. Limb amputation and limb deficiency: epidemiology and recent trends in the United States. South Med J. 2002 Aug;95(8):875-83. doi: 10.1097/00007611-200208000-00018. PMID 12190225